CLINICAL TRIAL: NCT06279715
Title: Evaluation of the Association Between the DNA Fragmentation Index (DFI) and the Frequency of Segmental and Total Aneuploidies
Brief Title: DFI and Aneuploidies
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3437
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-02

CONDITIONS: Embryo Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Preimplantation Genetic Testing for Aneuploidy — PGT-A typically involves the biopsy of three to eight cells from the developing embryo after approximately five days of culture. This technology also allows for the identification of segmentally aneuploid embryos.

SUMMARY:
IVF is the most commonly employed form of assisted reproductive technologies (ART) for the 10-15% of couples who face difficulties becoming pregnant. Many individuals elect to have their IVF-derived embryos analyzed using pregenetic implantation testing for aneuploidies (PGT-A). The use of PGT-A is particularly beneficial for patients at higher risk for aneuploidy, such as those of advanced maternal age and those faced with recurrent pregnancy loss or recurrent implantation failure.

Segmental aneuploidies are generated when a small piece of a chromosome is gained or lost during cell division, resulting in subchromosomal copy number (CN) changes. The frequency of segmental aneuploidies during the cleavage stage varies between studies, from as low as 3.9% to 15% and up to 70 % with no reported correlation with maternal age. This can be explained by the fact that, unlike whole chromosome aneuploidies, segmental aneuploidies most often involve paternally inherited chromosomes.

ELIGIBILITY:
Inclusion Criteria:

* IVF cycle completed at clinique ovo
* Maternal age between 18 to 43 years included
* PGT-A done on all embryos
* Recent DFI within 1 year of the IVF cycle

Exclusion Criteria:

* Sperm donation

Ages: 18 Years to 43 Years | Sex: All
Age Groups: Adult
Study Population: Data spreadsheet from October 2020 to December 2023 consisting of more than 800 medical charts.
Sampling Method: Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
DFI association and aneuploidy | Up to 3 weeks after embryo fertilization
  Segmental aneuploidy is associated with high levels of sperm DNA fragmentation index

CONTACTS AND LOCATIONS:
Overall Officials: Isaac-Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No